CLINICAL TRIAL: NCT01654731
Title: Multicenter, Randomized, Double-blind Placebo Controlled Trial of Bezafibrate for the Treatment of Primary Biliary Cirrhosis in Patients With Incomplete Response to Ursodesoxycholic Acid Therapy.
Brief Title: Phase 3 Study of Bezafibrate in Combination With Ursodeoxycholic Acid in Primary Biliary Cirrhosis
Acronym: BEZURSO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P100109; AOM 10291 (Other: Assistance Publique)
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: PBC
Keywords: PBC; Bezafibrate
MeSH Terms: interventions — Bezafibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bezafibrate (Experimental): 400 mg/Day
  Interventions: Drug: Bezafibrate
- Placebo (Placebo Comparator): 1 tablet/ day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Bezafibrate
  Arms: Bezafibrate
Drug: placebo
  Arms: Placebo

SUMMARY:
Primary biliary cirrhosis (PBC) is a chronic cholestatic liver disease that eventually leads to end-stage liver failure and death unless liver transplantation (LT) is performed. Ursodeoxycholic acid (UDCA) administered orally at the daily dose of 13-15 mg/kg is currently the only drug approved for the treatment of PBC. UDCA consistently improves biochemical liver tests, prolongs survival without LT, and delays histological progression as well as the occurrence of portal hypertension. However, a significant proportion (40%) of patients treated with UDCA shows an incomplete biochemical response and remains at high risk of death or LT. The development of new treatments in combination with UDCA is therefore needed. Several candidates exist among which is Bezafibrate. Bezafibrate belongs to the fibrates' pharmacological class, which has been developed 4 decades ago for the treatment of mixed hyperlipidaemia. Bezafibrate is cheap, widely available and well tolerated. There is now a substantial body of circumstantial evidence supporting that fibrates, and Bezafibrate in particular, are well tolerated and can improve biochemical liver tests in patients with PBC with incomplete response to UDCA. However, despite several positive successful pilot studies, there are still no phase 3 randomized placebo-controlled trials of fibrates for the treatment of PBC. The purpose of this protocol is therefore to conduct such a trial in a selected population of patients with PBC based on an incomplete biochemical response after 6 months of UDCA therapy.

DETAILED DESCRIPTION:
This is a multi-center, randomized (treatment will be assigned by chance), placebo-controlled (an inactive substance will be compared with the test drug to see whether the drug has a real effect), parallel-group (two or more groups of patients will receive different treatments) study that will assess the efficacy and safety of bezafibrate in patients with primary biliary cirrhosis (PBC) who had an inadequate biochemical response to ursodeoxycholic acid, as defined by the Paris II criteria. Bezafibrate 400 mg or placebo will be daily administered in combination with ursodeoxycholic acid (UDCA) 13-15 mg/kg/d for 24 months. Patient safety will be monitored. Primary end-point will be the percentage of patients with a complete normalization of the following biochemical tests: alkaline phosphatase, aminotransferases, total bilirubin, serum albumin, and prothrombin index. Secondary endpoints will include the percentage of drug-related adverse events, survival rates without liver transplantation or liver decompensation, time course of non-invasive liver fibrosis measurements (Fibroscan, serum hyaluronic acid), time course of liver histological parameters (fibrosis stage, necro-inflammatory grade, ductopenia) assessed on percutaneous biopsy specimens, time course of endoscopic, ultrasound, and biochemical features of portal hypertension, time course of pruritus and of quality of life using validated scales.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Patient with PBC defined by 2 in 3 of the following criteria Positive antimitochondrial antibody type M2. Abnormal serum alkaline phosphatases (ALP > 1,5N) and aminotransferase (AST or ALT > 1N) activities.

Histological hepatic injuries consistent with PBC from biopsy specimens of at least 10 mm.

* Patient treated with UDCA at the dose of 13 to 15 mg/kg/d (consistent to the AMM)
* Patients showing an incomplete biochemical response to UDCA as defined by : ALP > 1,5N or AST > 1,5N or total bilirubin >17 µmol/l (with conjugated bilirubin > 8 µmol/l) after ≥ 3 months of UDCA at the dose of 13 - 15 mg/kg/day.

Exclusion Criteria:

* Unsigned consent.
* Patient with no social insurance or having medical assistant of state
* Ascites or gastrointestinal bleeding (or history of these)
* Serum total bilirubinemia > 50 μmols/L (3 mg/dl) (sample < 3 months)
* Serum albuminemia < 35 g/l (sample < 3 months)
* Prothrombin index < 70% (sample < 3 months)
* Platelet count < 100000/mm3 (sample < 3 months)
* Treatment with corticosteroids, immunosuppressive agents, fibrates (or other PPAR-agonists) or statin in the last 3 months
* Any comorbidity susceptible to cause a hepatic impairment (HBV, HCV, or HIV seropositivity; excessive alcohol consumption; hemochromatosis, Wilson's disease, α1 antitrypsin deficiency; celiac disease; uncontrolled dysthyroidism; autoimmune hepatitis, inflammatory colitis)
* Any severe comorbidity decreasing life expectancy
* Intolerance or hypersensitivity to fibrates, to one of these components or other fibrates in general
* Known photosensitivity reaction to fibrates
* Pregnancy or desire of pregnancy
* Breast-feeding
* Renal failure (clearance of creatinine < 60 ml/mn)
* Patient with congenital galactosemia, syndrome of glucose malabsorption, lactase deficiency due to the presence of lactose in tablets of bezafibrate 400 mg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-10-15 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with complete biochemical response. | 24 months
  The normalisation of hepatic biochemical tests (aminotransferases (AST, ALT), Alkaline Phosphatase, blood Albumin, blood bilirubin and prothrombin index).

SECONDARY OUTCOMES:
Percentage of patients having biological or clinical adverse reaction. | 24 months
  Increase of ALT, AST or CPK > 5N
Percentage of patients having complete biochemical response. | 12 months
  Percentage of patients having complete biochemical response at Month 12.
Evolution of the pruritus. | 24 months
  Pruritus is measured via visual analogical scale every 3 months from month 0 to month 24
Assessment of the fatigue and the quality of life. | 24 months
  Measured via French questionnaire version of NHP (Nottingham Health Profile) every 12 months from month 0 to month 24
Evolution of liver fibrosis surrogate markers. | 24 months
  assessment of hyaluronic acid serum concentration and hepatic transient elastography (Fibroscan®)
Evolution of the portal hypertension markers. | 24 months
  Occurrence of ascites, decrease in the platelet count below 150000/mm3 or of more than 30% of its initial value, evolution of the ultrasound data of the splanchnic circulation, occurrence or size progression of oesophageal varices (endoscopy)
Histological evolution: Histopathological examination of biological sample before enrolment and at the end of the study. | 24 months
  Quantification of the fibrosis and the inflammatory and destructive injuries.
Evolution of the biological markers of the hepatic function or being in the usual prognostic scores (Mayo, Child, MELD). | 24 months
  Blood albumin, prothrombin time, INR, blood bilirubin, creatinine blood level.
Survival without transplantation and hepatic impairment. | 24 months
  Occurrence of ascites, a digestive variceal bleeding, a hepatic encephalopathy, or a doubling of the total blood bilirubin exceeding the threshold of 50 µmols/L (3 mg/dl).

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Corpechot, Doctor, Principal Investigator — Assistance Publique
Locations (1):
- Hepatology department - Hopital Saint Antoine, Paris, France

REFERENCES:
- [Background] Corpechot C, Chazouilleres O, Rousseau A, Le Gruyer A, Habersetzer F, Mathurin P, Goria O, Potier P, Minello A, Silvain C, Abergel A, Debette-Gratien M, Larrey D, Roux O, Bronowicki JP, Boursier J, de Ledinghen V, Heurgue-Berlot A, Nguyen-Khac E, Zoulim F, Ollivier-Hourmand I, Zarski JP, Nkontchou G, Lemoinne S, Humbert L, Rainteau D, Lefevre G, de Chaisemartin L, Chollet-Martin S, Gaouar F, Admane FH, Simon T, Poupon R. A Placebo-Controlled Trial of Bezafibrate in Primary Biliary Cholangitis. N Engl J Med. 2018 Jun 7;378(23):2171-2181. doi: 10.1056/NEJMoa1714519. PMID 29874528
- [Derived] Corpechot C, Chazouilleres O, Lemoinne S, Rousseau A. Letter: reduction in projected mortality or need for liver transplantation associated with bezafibrate add-on in primary biliary cholangitis with incomplete UDCA response. Aliment Pharmacol Ther. 2019 Jan;49(2):236-238. doi: 10.1111/apt.15049. No abstract available. PMID 30589964
- See also: Results — https://pubmed.ncbi.nlm.nih.gov/29874528/